CLINICAL TRIAL: NCT06934512
Title: Clinical Comparison of Pain Score of Needleless Jet Injector and Conventional Needle Injection for Teeth Extraction Anesthesia (Split Mouth Technique).
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Zahra Iftikhar, Principal Investigator Dr. Zehra Iftikhar, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-3820/DUHS/Approval/2025/73
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Pain Score
Keywords: Pain score

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Needleless jet injector (Experimental): Local anesthesia with needleless jet injector will be given on one site for the tooth extraction
  Interventions: Device: Needleless jet injector
- Conventional needle injection (Experimental): Local anesthesia with traditional needle will be given on another site for the tooth extraction
  Interventions: Procedure: Conventional needle injection

INTERVENTIONS:
Device: Needleless jet injector — To assess the pain score through (VAS) scale of needleless jet injector for local anesthesia. Scale has minimum zero number that indicates best outcome and maximum number is ten that indicates worst outcome.
  Arms: Needleless jet injector
Procedure: Conventional needle injection — To assess the pain score through (VAS) scale of traditional needle injection for local anesthesia. Scale has minimum zero number that indicates best outcome and maximum number is ten that indicates worst outcome.
  Arms: Conventional needle injection

SUMMARY:
Dental anesthesia with needle injection cause fear and anxiety in patients about the dental procedures. Therefore, less painful anesthesia alternatives like needleless anesthesia devices to reduce the negative sensation of pain and fear that is always associated with traditional local anesthesia needle injection.

The jet injector with INJEX is a needleless injector system that injects the local anesthesia solution into the tissues through a pressure. This research aims to compare the pain score of jet injector with INJEX and traditional local anesthesia needle injection for teeth extraction.

Method:

50 patients visiting DOW Ojha Hospital, who needs extraction of bilateral teeth will be included in this study. Data collection approval will be taken from Institutional Review Board (IRB) of DUHS.

Complete procedure, study purpose and pain scale will be explained to patients and they will be told that information will be utilized for only research purpose and after that permission will be taken from participants.

After taking history, quadrants will be divided; one for local anesthesia by the Jet Injector with INJEX and one for traditional local anesthesia needle injection.

After that local anesthesia with Jet Injector INJEX will be given to one side and traditional local anesthesia needle injection will be given to other site for teeth extraction. Then principle investigator will examine the patient pain through the pain scale (Visual Analog Scale) of this study and supervisor will confirm it.

ELIGIBILITY:
INCLUSION CRITERIA:

* 18-24 years old patient
* Patients having permanent dentition who require bilateral anterior or premolar teeth extraction
* Orthodontic patients who requires bilateral extraction of premolars
* Patients who give informed consent to take part in study

EXCLUSION CRITERIA:

* Patients with local anesthesia allergy
* Patients with localized inflammation/ localized abscess/tenderness at site of injection
* Patients who do not give informed consent to take part in study

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
CLINICAL COMPARISON OF PAIN SCORE OF NEEDLELESS JET INJECTOR AND CONVENTIONAL NEEDLE INJECTION FOR TEETH EXTRACTION ANESTHESIA (SPLIT MOUTH TECHNIQUE) | Peri operative

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Dr. Ishrat-ul-Ebad Institute of Oral Health Sciences, Karachi, Sindh
  - Dow University of Health and Sciences, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: No